CLINICAL TRIAL: NCT04538066
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Assessing Safety, Tolerability and Long-term Efficacy of Bryostatin in the Treatment of Moderately Severe Alzheimer's Disease Subjects Not Receiving Memantine Treatment
Brief Title: Bryostatin Treatment of Moderately Severe Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotrope Bioscience, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRP101-204; R44AG066366 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-09-03 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bryostatin 1

STUDY DESIGN:
Intervention Model Description: Study subjects will be randomized 1:1 to receive either the active treatment, bryostatin-1, or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, investigators and staff, and the clinical research organization are all blinded to study treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bryostatin 1 (Active Comparator): 20ug Bryostatin will be administered over 45 minutes IV. The course of treatment will include 7 doses over the first 12 weeks, followed by a second identical treatment period beginning 30 days after completion of the first treatment period.
  Interventions: Drug: Bryostatin 1
- Placebo (Placebo Comparator): Placebo will be administered over 45 minutes IV. The course of treatment will include 7 doses over the first 12 weeks, followed by a second identical treatment period beginning 30 days after completion of the first treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bryostatin 1 — Bryostatin 20 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks, followed by a second identical course of treatment beginning 30 days after completion of the first 7-dose course.
  Arms: Bryostatin 1
Other: Placebo — Placebo administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks, followed by a second identical course of treatment beginning 30 days after completion of the first 7-dose course.
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability, and long-term efficacy of bryostatin 1 (hereafter referred to as bryostatin) for the treatment of moderately severe Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled, Phase 2 study comparing bryostatin-1 to placebo for long-term efficacy in the treatment of moderately severe AD (Mini Mental State Examination, 2nd edition scores of 10-18 at baseline) in the absence of memantine. Eligible subjects will receive 7 doses of bryostatin (i.v., 20μg) or matching placebo during the first 12 weeks. A second course of treatment consisting of 7 doses will begin 30 days after the final dose of the first treatment period. Cognitive tests will be assessed at intervals during the study and 4 months after the final dose of study drug. The primary endpoint is the total SIB score assessment obtained at Week 28, following completion of 2 courses of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from caregiver and subject (if possible) or legally acceptable representative if different from caregiver
2. Male and female subjects 55-85 years of age inclusive
3. Cognitive deficit present for at least 2 years that meet the diagnostic criteria for probable Alzheimer's dementia. The diagnosis must be confirmed at the time of the screening visit
4. MMSE-2 score of 10-18 inclusive (applies to Screening Visit only)
5. Patients must have a baseline SIB total score of at least 60 and may not have a SIB score >93 at screening
6. Neuroimaging computerized tomography (CT) or Magnetic Resonance Imaging (MRI) within the last 24 months consistent with a diagnosis of probable AD without any other clinically significant co-morbid pathologies. If there has been a significant change in the subject's clinical status since the last imaging study that is not consistent with progression of the subject's AD, an imaging study should be performed to confirm eligibility
7. Reliable caregiver(s) or informant(s) who attends the subject at least an average of 3 hours or more per day for 3 or more days per week and who will agree to accompany the subject to the clinic visits and reliably complete the caregiver questions
8. Adequate vision and motor function to comply with testing
9. If taking an approved cholinesterase inhibitor for treatment of Alzheimer's disease, must be on a stable dose for at least 3 months prior to entry into study and the dose must not change during the study unless a change is required due to an adverse effect of the prescribed medication or a clinically significant change in the patient's status
10. Subjects who are memantine naïve or have been off memantine for at least 90 days prior to initial treatment with study drug
11. Subjects on neuroleptic medications must be on a stable dose for ≥4 weeks at screening (dose adjustments will be permitted if medically necessary at the discretion of the PI)
12. Females participating in the study must meet one the following criteria:

    1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
    2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) 30 days prior to dosing until 30 days after last dose and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at screening
13. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) from 30 days prior to dosing until 30 days after last dose
14. In the opinion of the PI subjects should be in reasonably good health over the last 6 months and any chronic disease should be stable -

Exclusion Criteria:

Eligibility Criteria:

Inclusion

1. Written informed consent from caregiver and subject (if possible) or legally acceptable representative if different from caregiver 2. Male and female subjects 55-85 years of age inclusive 3. Cognitive deficit present for at least 2 years that meet the diagnostic criteria for probable Alzheimer's dementia. The diagnosis must be confirmed at the time of the screening visit 4. MMSE-2 score of 10-18 inclusive (applies to Screening Visit only) 5. Patients must have a baseline SIB total score of at least 60 and may not have a SIB score >93 at screening 6. Neuroimaging computerized tomography (CT) or Magnetic Resonance Imaging (MRI) within the last 24 months consistent with a diagnosis of probable AD without any other clinically significant co-morbid pathologies. If there has been a significant change in the subject's clinical status since the last imaging study that is not consistent with progression of the subject's AD, an imaging study should be performed to confirm eligibility 7. Reliable caregiver(s) or informant(s) who attends the subject at least an average of 3 hours or more per day for 3 or more days per week and who will agree to accompany the subject to the clinic visits and reliably complete the caregiver questions 8. Adequate vision and motor function to comply with testing 9. If taking an approved cholinesterase inhibitor for treatment of Alzheimer's disease, must be on a stable dose for at least 3 months prior to entry into study and the dose must not change during the study unless a change is required due to an adverse effect of the prescribed medication or a clinically significant change in the patient's status 10. Subjects who are memantine naïve or have been off memantine for at least 90 days prior to initial treatment with study drug 11. Subjects on neuroleptic medications must be on a stable dose for ≥4 weeks at screening (dose adjustments will be permitted if medically necessary at the discretion of the PI) 12. Females participating in the study must meet one the following criteria:

1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) 30 days prior to dosing until 30 days after last dose and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at screening 13. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) from 30 days prior to dosing until 30 days after last dose 14. In the opinion of the PI subjects should be in reasonably good health over the last 6 months and any chronic disease should be stable Exclusion

   1. Dementia due to any condition other than AD, including vascular dementia (Rosen-Modified Hachinski Ischemic score ≥ 5)
   2. Evidence of significant central nervous system (CNS) vascular disease on previous neuroimaging including but not limited to: cortical stroke, multiple infarcts, localized single infarcts in the thalamus, angular gyrus, multiple lacunar infarcts or extensive white matter injury
   3. Clinically significant neurologic disease or condition other than AD, such as cerebral tumor, chronic subdural fluid collections, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, or any other diagnosis that could interfere with assessment of safety and efficacy
   4. Evidence of clinically significant unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurologic, or metabolic disease within the 6 months prior to enrollment. If there is a history of cancer the subject should be clear of cancer for at least 2 years prior to screening. More recent history of basal cell or squamous cell carcinoma and melanoma in situ (Stage 0) may be acceptable after review by the Medical Monitor.
   5. Creatinine clearance (CL) of <45ml/min
   6. Poorly controlled diabetes, at the discretion of the Principal Investigator
   7. Concomitant treatment with NMDA receptor antagonists such as but not limited to memantine or drug combinations containing memantine, dextromethorphan (a cough suppressant), ketamine, phencyclidine (PCP), methoxetamine (MXE), nitrous oxide (N2O) and the following synthetic opioids: penthidine, levorphanol, methadone, dextrpropoxyphene, tramadol, and ketobemidone.
   8. Use of vitamin E > 400 International Units (IU) per day within 14 days prior to screening
   9. Use of acetaminophen within 14 days prior to screening
   10. Use of gabapentin within 14 days prior to screening
   11. Use of valproic acid within 14 days prior to screening
   12. Use of an active Alzheimer's vaccine within 2 years prior to screening
   13. Use of a monoclonal antibody for treatment of AD within 1 year prior to screening
   14. Any medical or psychiatric condition that is likely to require initiation of additional medication or surgical intervention during the course of the study
   15. Any screening laboratory values outside the reference ranges that are deemed clinically significant by the PI
   16. Use of an investigational drug within 90 days prior to screening
   17. Suicidality defined as active suicidal thoughts during the 6 months prior to screening or at Baseline [Type 4 or 5 on C-SSRS], or history of suicide attempt in previous 2 years, or at serious suicide risk in PI's judgment
   18. Major psychiatric illness such as current major depression according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition , current or past diagnosis of bipolar disorder, schizophrenia, or any other psychiatric disorder that might interfere with the assessments of safety or efficacy at the discretion of the PI
   19. Diagnosis of alcohol or drug abuse within the last 2 years
   20. Abnormal laboratory tests that suggest an alternate etiology for dementia. If the patient has prior history of serum B12 abnormality, anemia with hemoglobin ≤10g/dl, thyroid function abnormality, electrolyte abnormality, or positive syphilis serology the patient should be revaluated to determine if these potential causes of dementia have been addressed. Only if these causes have been ruled out as the cause of the dementia can the patient be enrolled.
   21. History of prolonged QT or prolonged QT on screening ECG (QTcB or QTcF >499 per central reader)
   22. Acute or poorly controlled medical illness: blood pressure > 180 mmHg systolic or 100 mmHg diastolic; myocardial infarction within 6 months; uncompensated congestive heart failure [New York Heart Association (NYHA) Class III or IV]
   23. Known to be seropositive for human immunodeficiency virus (HIV)
   24. Known to be seropositive for Hepatitis B or C, unless successful curative treatment for Hepatitis C (e.g., Harvoni) has been received and there is documentation that there is no Hep B/C virus detected 3 months after completion of treatment
   25. AST or ALT >3x upper limit of normal (ULN) and total bilirubin >2x ULN or International Normalized Ratio (INR) >1.5
   26. Prior exposure to bryostatin, or known sensitivity to bryostatin or any ingredient in the study drug
   27. Any other concurrent medical condition, which in the opinion of the PI makes the subject unsuitable for the clinical study -

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Axiom Research, Colton, California
  - Pacific Research Network, San Diego, California
  - JEM Research, Atlantis, Florida
  - Galiz Research, Hialeah, Florida
  - ClinCloud, Maitland, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Columbus Memory Center, Columbus, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Millenium Psychiatric Associates, St Louis, Missouri
  - Neurological Associates of Albany, P. C., Albany, New York
  - Alzheimer's Research Center, Matthews, North Carolina
  - Summitt Research Network (Oregon), Portland, Oregon
  - Kingfisher Cooperative, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine medical clinics in the US were selected to recruit study subjects.
Period: Overall Study
Arm/Group | Bryostatin 1 | Placebo
Started (Although 122 subjects were randomized, only 117 proceeded to participate.) | 61 | 61
Completed | 33 | 40
Not Completed | 28 | 21

BASELINE CHARACTERISTICS:
Population: Although 61 subjects in each arm were randomized and assigned to either receive bryostatin or placebo, 5 subjects were never dosed, bringing the number of subjects who received treatment to 59 bryostatin and 58 placebo (117 total).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bryostatin 1 | Placebo | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 52 | 48 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (7.64) | 73.1 (7.69) | 73.9 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 32 | 30 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 52 | 53 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 117
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.53 (4.691) | 26.89 (4.119) | 26.71 (4.401)

OUTCOME MEASURES:

1. Primary Outcome: Safety: Treatment-emergent Adverse Events and Serious Adverse Events for All Randomized Subjects Who Received Any Study Medication
Description: Treatment emergent adverse events and serious adverse events will be analyzed by treatment group.
Time Frame: Prior to version 6 of the protocol, final assessments were performed at Week 42, 12 weeks after the last study treatment. The final study visit took place at Week 30 for subjects remaining in the study after the protocol amendment.
Population: All subjected who received any dose of study drug were included in the safety analysis.
Measure: Number; unit: number of events
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 59 | 58
number of events
  Treatment related treatment emergent adverse event (TEAE) | 15 | 13
  Serious TEAE | 4 | 4
  TEAE leading to early discontinuation of study treatment | 6 | 6
  TEAE leading to study termination | 3 | 3

2. Primary Outcome: Efficacy: Severe Impairment Battery Total Score Assessment Obtained After Completion of the Second Couse of Treatment (Week 28)
Description: The treatment difference in the primary efficacy endpoint of Severe Impairment Battery (SIB). The SIB is used to assess cognition in subjects with moderate and severe AD. It is divided into nine subscales that include attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Primary efficacy analysis at Week 28
Population: All subjects who completed Week 28 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 31 | 34
score on a scale | 1.7 (1.44) | 0.2 (1.46)

3. Secondary Outcome: Severe Impairment Battery (SIB) Total Score at the End of the Week 42 Follow-up Visit
Description: The SIB assesses cognition. Score range 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Week 42 was the final follow-up for study subjects, occurring 16 weeks after the last dose of study drug. Subjects who remained in the study at the time version 6 of the protocol was implemented did not have Week 42 visit.
Population: All subjects who completed Week 42 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 28 | 36
score on a scale | 88.4 (1.81) | 84.3 (1.59)

4. Secondary Outcome: The SIB Total Score From Baseline at Week 13
Description: The SIB assesses cognition. Score range 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Week 13 followed the first 12-week course of study treatment.
Population: All subjects who completed Week 13 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 49 | 49
score on a scale | 2.4 (0.87) | 1.7 (0.87)

5. Secondary Outcome: The Changes From Baseline in SIB Total Scores at Weeks 9, 20, 24, and 30
Description: The Severe Impaorment Battery (SIB) assesses cognition. Score range 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Weeks 9, 20 and 24 occur during the treatment phase of the study. Week 30 occurred 4 weeks after end of treatment.
Population: All subjects who completed Week 9 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 43 | 46
score on a scale
  Week 9 | 1.9 (0.77) | 1.3 (0.80)
  Week 20: number analyzed (Participants) | 37 | 39
  Week 20 | 1.8 (1.09) | 0.7 (1.11)
  Week 24: number analyzed (Participants) | 30 | 37
  Week 24 | 1.7 (1.26) | 0.4 (1.27)
  Week 30 | 1.7 (1.54) | 0.1 (1.55)

6. Secondary Outcome: SIB Total Scores From Baseline at Weeks 9, 20, 24 and 30 for Subjects With Baseline Mini Mental State Exam Version 2 (MMSE-2) Scores of 10-14 and 15-18
Description: MMSE-2 tests selected aspects of cognition on a scale of 0-30. Subjects with MMSE-2 scores of 10-18 will be enrolled in the study. Scores of 10-14 indicate greater impairment than scores of 15-18. Analyses were done comparing all subjects treated with either bryostatin or placebo, and additionally, comparing subjects grouped by MMSE-2 scores of 10-14 and 15-18 treated with either bryostatin or placebo.
Time Frame: Weeks 9, 20, 24 and 30
Population: The decline in number of participants analyzed reflects attrition in number of subjects remaining in the trial at each successive timepoint.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Bryostatin Baseline MMSE-2 Score 10 to 14; Placebo Baseline MMSE-2 Score 10-14: Subjects with MMSE-2 score of 10-14 at Baseline. The MMSE-2 measures selected aspects of cognition such as memory, orientation, attention, language, and praxis on a scale of 0 to 30. Lower scores indicate greater cognitive impairment than higher scores.
- Bryostatin Baseline MMSE-2 Score 15-18; Placebo Baseline MMSE-2 Score 15-18: Subjects with MMSE-2 score of 15-18 at Baseline. The MMSE-2 measures selected aspects of cognition such as memory, orientation, attention, language, and praxis on a scale of 0 to 30. Lower scores indicate greater cognitive impairment than higher scores.
Arm/Group | Bryostatin Baseline MMSE-2 Score 10 to 14 | Placebo Baseline MMSE-2 Score 10-14 | Bryostatin Baseline MMSE-2 Score 15-18 | Placebo Baseline MMSE-2 Score 15-18
Number analyzed (Participants) | 25 | 27 | 25 | 24
scores on a scale
  Week 9: number analyzed (Participants) | 18 | 22 | 25 | 24
  Week 9 | 0.8 (1.37) | -2.6 (1.32) | 3.3 (0.61) | 4.5 (0.66)
  Week 20: number analyzed (Participants) | 16 | 19 | 21 | 20
  Week 20 | 0.1 (1.87) | -5.6 (1.81) | 3.9 (0.60) | 5.5 (0.62)
  Week 24: number analyzed (Participants) | 11 | 18 | 19 | 19
  Week 24 | -0.1 (2.18) | -6.7 (2.11) | 4.1 (0.66) | 5.8 (0.67)
  Week 30: number analyzed (Participants) | 11 | 15 | 14 | 21
  Week 30 | -0.4 (2.70) | -8.3 (2.62) | 4.4 (0.79) | 6.3 (0.78)

7. Secondary Outcome: SIB Trends Over Time
Description: Individual-specific slopes of total Severe Impairment Battery (SIB) scores will be obtained for all patients. Scores range from 0-100, lower scores indicate greater impairment.
Time Frame: Slopes will be estimated by using SIB data at Week 0, 5, 9, 13, 15, 20, 24, and 28
Population: All subjects who received any dose of study drug were included in the full analysis set (FAS), 117 subjects.
Measure: Mean (95% Confidence Interval); unit: scores on a scale / week, averaged for e
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 57 | 55
scores on a scale / week, averaged for e | -1.2863 [-2.0944 to -0.4782] | -1.3205 [-2.1226 to -0.5184]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from 8/19/2020 (first subject screened) to 11/16/22 (last subject follow-up visit). Prior to the version 6 amendment to the study protocol, adverse events were also collected from participants at week 42, 16 weeks after last dose. After the amendment, adverse events were collected up to week 30, the final study visit, or 30 days after the last dose.
Description: Subjects' adverse events were recorded from the date of screening until 30 days after the last study drug dose.
Arm/Group | Bryostatin 1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 3/59 | 3/58
Other Adverse Events (participants affected / at risk) | 35/59 | 30/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 1 (N=59) | Placebo (N=58)
colon tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
fractured vertebrae (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fractured R femur (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
macrocytic anemia d/t B-12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
acute metabolic encephalopathy (General disorders) | 1 (1) | 0 (0)
altered mental state (Nervous system disorders) | 1 (1) | 0 (0)
colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 1 (N=59) | Placebo (N=58)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (8) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
General disorders and administrative site conditions (General disorders) | 5 (6) | 3 (3)
Infusion site extravasation (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Infections and infestations (Infections and infestations) | 9 (13) | 14 (16)
Covid-19 (Infections and infestations) | 4 (4) | 0 (0)
Sinusitis (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (4)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (4) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Investigations (Investigations) | 5 (5) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Nervous system disorders (Nervous system disorders) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 8 (10) | 8 (14)
Agitation (Psychiatric disorders) | 5 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Hallucination (Psychiatric disorders) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Vascular disorders (Vascular disorders) | 4 (4) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Phlebitis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to the primary publication. Following primary publication, the PI may publish results from the Study but must submit the publication to Sponsor for approval at least 60 days prior to journal submission. If there is patentable subject matter in the proposed publication, publication shall be delayed to allow for the preparation of a patent application. If primary manuscript is not submitted within 12 months after end of the Study, PI may publish own Study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04538066/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04538066/SAP_001.pdf